CLINICAL TRIAL: NCT02171962
Title: Evaluation of the Zilver® PTX® Drug-Eluting Peripheral Stent for Treatment of Lesions of the Above-the-Knee Femoropopliteal Artery
Brief Title: Zilver® PTX® in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-008
Record Dates: First submitted 2014-06-18; First posted 2014-06-24 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Peripheral Artery Disease
Keywords: Zilver® PTX® Drug-Eluting Peripheral Stent; Above-the-Knee Femoropopliteal Artery; Chinese patient
MeSH Terms: conditions — Peripheral Arterial Disease

ARMS (1):
- Zilver® PTX® VI (Experimental)
  Interventions: Device: Zilver® PTX® Drug-Eluting Peripheral Stent

INTERVENTIONS:
Device: Zilver® PTX® Drug-Eluting Peripheral Stent — Zilver® PTX® Drug-Eluting Peripheral Stent for treatment of lesions of the above-the-knee femoropopliteal artery

SUMMARY:
The objective of this study is to evaluate the Zilver® PTX® Drug-Eluting Peripheral Stent for treatment of lesions of the above-the-knee femoropopliteal artery in a Chinese patient population.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of peripheral arterial disease corresponding to Rutherford Classification 2-4
* Stenotic (>50% diameter stenosis) or occluded lesion of the above-the knee femoropopliteal artery
* Reference vessel diameter of 4-9 mm
* Lesion length up to 140 mm

Exclusion Criteria:

* Unsuccessful arterial interventional treatment of the legs within 30 days prior to the study procedure
* Previous stent in the study vessel
* Bypass graft with an anastomosis in the study vessel
* Significant stenosis or occlusion of inflow tract not successfully treated prior to treating the study lesion
* No patent vessel of runoff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2017-02-09 (Actual)

PRIMARY OUTCOMES:
Primary Patency as Assessed by Duplex Ultrasonography | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dake, MD, Study Director — Stanford University, CA, USA; Changwei Liu, MD, Principal Investigator — Peking Union Medical College Hospital, Beijing, China; Weiguo Fu, MD, Principal Investigator — Zhongshan Hospital Fudan University, Shanghai, China
Locations (9):
- China (9):
  - Beijing Anzhen Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Shanghai Ninth People's Hospital Affiliated Shanghai JiaoTong University School of Medicine, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai

REFERENCES:
- [Derived] Ye W, Bohme T, Fu W, Liu C, Zhang X, Liu P, Zhang J, Zou Y, Lu X, Lottes AE, O'Leary EE, Zeller T, Dake MD. First peripheral drug-eluting stent clinical results from China: 1-year outcomes of the Zilver PTX China study. Front Cardiovasc Med. 2022 Sep 27;9:877578. doi: 10.3389/fcvm.2022.877578. eCollection 2022. PMID 36237908
- [Derived] Dake MD, Fanelli F, Lottes AE, O'Leary EE, Reichert H, Jiang X, Fu W, Iida O, Zen K, Schermerhorn M, Zeller T, Ansel GM. Prediction Model for Freedom from TLR from a Multi-study Analysis of Long-Term Results with the Zilver PTX Drug-Eluting Peripheral Stent. Cardiovasc Intervent Radiol. 2021 Feb;44(2):196-206. doi: 10.1007/s00270-020-02648-6. Epub 2020 Oct 6. PMID 33025243